CLINICAL TRIAL: NCT02096952
Title: Open-Label Treatment Trial to Assess the Short-Term Tolerability, Safety, and Efficacy of Methylphenidate Hydrochloride Extended-Release Liquid Formulation in High-Functioning Autism Spectrum Disorder Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: Methylphenidate ER Liquid Formulation in Adults With ASD and ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Assistant professor of Psychiatry, Harvard Medical School; Director, Autism Spectrum Disorder Clinical & Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000501
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Attention-deficit/Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: Attention-deficit/hyperactivity disorder; ADHD; Autism spectrum disorder; ASD; High-functioning ASD; Asperger's disorder; Asperger's
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Asperger Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylphenidate extended-release liquid (Experimental): Methylphenidate extended-release liquid formulation
  Interventions: Drug: Methylphenidate extended-release liquid formulation

INTERVENTIONS:
Drug: Methylphenidate extended-release liquid formulation
  Other Names: Quillivant extended release

SUMMARY:
The purpose of this study is to determine whether methylphenidate hydrochloride extended release liquid formulation is safe and effective in the treatment of attention-deficit/hyperactivity disorder (ADHD) in high-functioning adults with autism spectrum disorders (ASD).

ELIGIBILITY:
Inclusion Criteria

* Male or female participants between 18 and 40 years of age (inclusive)
* Fulfills DSM-5 diagnostic criteria for autism spectrum disorder as established by the clinical diagnostic interview and ADOS
* Fulfills DSM-5 diagnostic criteria for ADHD as established by the clinical diagnostic interview and confirmed by the K-SADS-E ADHD module
* Participants with at least moderately severe symptoms of ASD as demonstrated by SRS raw score ≥ 85 and CGI-ASD severity score ≥ 4
* Participants with at least moderately severe symptoms of ADHD as assessed by AISRS score ≥ 24 and CGI-ADHD severity score ≥ 4
* Participants and/or their legal representative must understand the nature of the study. Participants and/or their legal representative must sign an IRB-approved informed consent form before initiation of any study procedures.
* Participants and/or their legal representative must have a level of understanding sufficient to communicate with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Participant must be able to participate in mandatory blood draws.
* Participant with major mood and/or anxiety disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion Criteria

* Impaired intellectual capacity (IQ <85)
* Participant is unable to communicate due to delay in, or total lack of, spoken language development (grossly impaired language skills)
* Clinically unstable psychiatric conditions or judged to be at serious safety risk to self (suicidal risk) or others (within past 30 days).
* Subjects currently (within past 30 days) experiencing significant features of anxiety, mood, or psychotic disorder as indicated by a >3 score on the disorder-specific Clinical Global Impression-Severity (CGI-S) clinician-rated scale.
* History of substance use (except nicotine or caffeine) within past 3 months (inclusive) or with urine drug screen positive for substances of abuse
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:
* Pregnant or nursing females or females with a positive beta-HCG pregnancy test.
* Uncorrected hypothyroidism or hyperthyroidism.
* History of non-febrile seizures within last 1 month without a clear and resolved etiology.
* History of renal or hepatic impairment.
* Glaucoma
* Tourette's syndrome and/or motor tics
* Serious, unstable systemic illness
* Personal history of cardiac disease or a family history of non-geriatric cardiac disease or death
* Clinically significant abnormal baseline laboratory values which include the following:
* Values more than 20% above the upper range of the laboratory standard for a basic metabolic screen.
* Systolic and diastolic blood pressure parameters above 140 and 90, respectively.
* Resting heart rate outside of 60-100 bpm.
* Abnormal ECG parameters defined as QTC> 460msec, QRS>120 msec, and/or PR>200 msec.
* ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
* Participant with a history of non-response to adequate trial of methylphenidate (therapeutic dose for an adequate duration) as determined by clinician.
* History of intolerance or an allergic reaction to methylphenidate.
* Current or recent treatment (within the past 30 days) with current stimulant class of anti-ADHD medications.
* Current treatment with monoamine oxidase inhibitors (MAOIs)
* Current treatment with a first- or second-generation antipsychotic medication on a dose that has not been stable for at least 4 weeks prior to baseline visit.
* Current treatment with a psychotropic medication on a dose that has not been stable for at least 4 weeks prior to baseline visit.
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild.

While stably treated or remitted hypertension is not exclusionary, any subject with a history of high blood pressure will be asked to obtain approval from their primary care physician certifying that their hypertension is stable and that they may safely begin stimulant therapy. Subjects will be informed of the cardiovascular risks of MPH, and any subject with a history of hypertension who is unwilling to consult with their current treater-or to grant study staff permission to consult with the subject's current treater-will be excluded because of the potential risks to subject safety. Per the FDA approved MPH-ERLF package insert, high blood pressure is not a contraindication of MPH therapy; however, due to the cardiovascular side effects, it is recommended that subjects with a history of high blood pressure be monitored carefully. Cardiovascular risk factors are carefully monitored throughout the study for all subjects by way of screening electrocardiograms and pulse/blood pressure readings at every office visit. Patients with current untreated hypertension are not eligible.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joshi G, DiSalvo M, Wozniak J, Ceranoglu TA, Yule A, Surman C, Fried R, Galdo M, Hoskova B, Belser A, Biederman J. A prospective open-label trial of long-acting liquid methylphenidate for the treatment of attention deficit/hyperactivity disorder in intellectually capable adults with autism spectrum disorder. World J Biol Psychiatry. 2020 Apr;21(4):274-290. doi: 10.1080/15622975.2019.1679392. Epub 2019 Dec 19. PMID 31607204

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylphenidate Extended-release Liquid: Methylphenidate extended-release liquid formulation (MPH-ERLF)
  The MPH-ERLF was titrated to the target daily dose during the first three weeks of the trial (dose optimization phase) based on a flexible titration schedule as well as tolerability per clinician judgement. Week 3 and onwards, subjects were maintained on maximum achieved dose with a one-time option to decrease the dose of the study medication to the next lowest available dose per clinician judgement based on tolerability.
Period: Overall Study
Arm/Group | Methylphenidate Extended-release Liquid
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Methylphenidate Extended-release Liquid
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult ADHD Investigator Symptom Report Scale (AISRS) Score
Description: The Adult ADHD Investigator Symptom Report Scale (AISRS) assesses each of the 18 individual symptoms of ADHD in DSM-IV on a Likert scale from 0 (not present) to 3 (severe), with a total possible score of 54.
  The change in AISRS score from baseline to endpoint (6 weeks) was calculated as the later time point score minus the earlier time point score.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Extended-release Liquid
Number analyzed (Participants) | 15
units on a scale | -22.8 (8.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire time that subjects were exposed to the study medication (6 weeks)
Arm/Group | Methylphenidate Extended-release Liquid
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Extended-release Liquid (N=15)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Extended-release Liquid (N=15)
Headache (General disorders) | 8 (21)
Insomnia (Psychiatric disorders) | 5 (11)
Anxiety (Psychiatric disorders) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 4 (11)
Difficulty falling asleep (General disorders) | 3 (5)
Irritability (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (5)
Fatigue (General disorders) | 2 (4)
Tachycardia (Cardiac disorders) | 2 (2)
High blood pressure (Blood and lymphatic system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Heart racing (Cardiac disorders) | 1 (2)
Chest pressure (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Depressed mood (Psychiatric disorders) | 1 (1)
Jittery and tense (Psychiatric disorders) | 1 (1)
Sweaty hands (Skin and subcutaneous tissue disorders) | 1 (1)
Flu (Infections and infestations) | 1 (1)
Toothache (Infections and infestations) | 1 (1)
Sinus issues (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02096952/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02096952/ICF_001.pdf